CLINICAL TRIAL: NCT01067950
Title: International, Multicenter, Prospective, Randomized, Parallel Group, Open Label Protocol to Evaluate Safety and Efficacy of Isolated Pancreas Transplantation Compared to Intensive Insulin Therapy in Type 1 Diabetic Patients With Overt Diabetic Nephropathy and Mildly Reduced Renal Function
Brief Title: Pancreas Allotransplantation for Diabetic Nephropathy and Mild Chronic REnal fAilure Stage Study
Acronym: PANCREAS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: General Director, Nantes University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD 09/5-J
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-03

CONDITIONS: Type 1 Diabetes
Keywords: isolated pancreas transplant; intensive insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isolated Pancreas Transplant (Experimental)
  Interventions: Procedure: Isolated Pancreas Transplant
- Intensive Insulin Therapy (Active Comparator)
  Interventions: Drug: Intensive Insulin Therapy

INTERVENTIONS:
Procedure: Isolated Pancreas Transplant
  Arms: Isolated Pancreas Transplant
Drug: Intensive Insulin Therapy
  Arms: Intensive Insulin Therapy

SUMMARY:
Current medical therapies are not able to prevent progression of established macroproteinuira (i.e. diabetic nephropathy) to end-stage renal failure in type 1 (insulin dependent) diabetic patients. In this setting, proteinuria is a major risk factor for mortality. Pancreas transplantation, on the contrary, can revert diabetic nephropathy and thereby prevent end-stage chronic renal failure, with theoretically lower risk of death as compared to current medical therapies.The main objective of this study is to assess superiority of isolated pancreas transplantation versus intensive exogenous insulin therapy in type 1 diabetic patients with overt diabetic nephropathy and mildly reduced renal function. The primary endpoint is a composite efficacy/failure end-point including: patient mortality and renal function impairment during 5 years in patients with badly controlled diabetes and nephropathy resisting to up-to-date nephroprotective therapies.Main secondary objectives are safety and efficacy of both regimens, including proteinuria and renal histology evaluation, metabolic control and quality of life, acute and chronic extrarenal complications of diabetes, pancreas survival and all risks related to the transplant procedure (anaesthesia, surgery and immunosuppression side-effects) and to the intensive insulin therapy management.

ELIGIBILITY:
Inclusion Criteria:

Patients will be enroled in this study if they meet all of the following criteria:

* Type 1 diabetic patient aged between 25 and 55 years at the time of randomisation.
* Fasting plasma C-peptide below 0.5 ng/ml.
* Badly controlled diabetes despite an optimized insulin regimen consisting in continuous subcutaneous insulin infusion (via an insulin pump) or in multiple daily injections of insulin
* Persistent 24-hour proteinuria above 300 mg/day (a mean from 3 samples) despite adapted anti-proteinuric therapy for at least 6 months.
* Cystatin C and/or Cr51-EDTA and/or DMSA-Tc scintigraphy measured glomerular filtration rate from 60 to 90 ml/min.
* No contraindication to pancreas transplant surgery
* Woman of childbearing potential must have a negative serum pregnancy test at enrolment and must agree to maintain effective birth control during first year of the study.
* Capable of understanding the purpose and risks of the study, fully informed and given written informed consent (signed Informed Consent has been obtained).
* Affiliated to national insurance.

Exclusion Criteria:

Patients will be excluded from participating if any of the following criteria apply:

* Patient with any type 2 diabetes and/or fasting plasma C-peptide above 0.5 ng/ml.
* Pregnant woman or breast-feeding mothers.
* Woman of childbearing potential unwilling to maintain effective birth control during first year of the study
* Second transplant recipient or recipient with a functional grafted organ.
* Proteinuria below 300 mg/day (a mean from 3 samples).
* Albuminemia less than 30 g/l.
* Cystatin C and/or Cr51-EDTA and/or DMSA-Tc scintigraphy measured glomerular filtration rate lower than 60 ml/min or higher than 90 ml/min.
* Presence of any documented non-diabetic systemic disease potentially affecting the kidney.
* Known allergy, hypersensibility or intolerance to any known insulin, to any of the recommended immunosuppressive agents of the study (Thymoglobulin, anti-lymphocyte serum Fresenius, tacrolimus, cyclosporin, mycophenolate mofetil, mycophenolic acid, corticosteroids etc), mocrolides antibiotics, or to any compound or excipient of all these products.
* Currently participating in another clinical trial and/or has taken an investigational drug within four weeks prior enrolment.
* Diagnosis of new-onset malignancy during 5 years before enrolment.
* Significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastrointestinal tract malabsorption or active peptic ulcer.
* Patient affected by active B hepatitis (HBsAg positive, HBeAg positive or HBV-DNA positive) or by active C hepatitis (HCVAb positive; HCV-RNA positive).
* Patient HIV positive.
* Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the investigator.
* Obesity (body mass index above than 30 kg/m2).
* Severe iliac vessel calcifications impeding surgery.
* Advanced coronary artery disease
* Left ventricular function less than 30%.
* Plasma blood leukocytes less than 2,000 /mm3 or higher than 15,000/mm3
* Plasma blood platelets less 60,000 /mm3 or higher than 500,000/mm3
* Psychological disorders influencing drug compliance.
* Unable, unwilling or unlikely to comply fully with the protocol or the visits scheduled.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2010-03

PRIMARY OUTCOMES:
The primary end-point is the 5-year evaluation of efficacy/failure rate, a composite end-point including: (i) patient mortality and (ii) renal function impairment | 5 years

SECONDARY OUTCOMES:
Secondary objectives are to evaluate and to compare the safety and the efficacy of the two treatments (IPT versus IIT). | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Diego CANTAROVICH, MD, PhD, Principal Investigator — Nantes University Hospital
Locations (7):
- University of Minnesota, Minneapolis, Minnesota, United States
- Albert Einstein Jewish Hospital, São Paulo, Brazil
- Diabetes Center - Institute for Clinical and Experimental Medicine, Prague, Czechia
- France (2):
  - Hôpital Edouard-Herriot - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier et Universitaire de Nantes, Nantes
- Italy (2):
  - Istituto Scientifico Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria Pisana, Pisa